CLINICAL TRIAL: NCT07288164
Title: Comparison of Operative and Early Postoperative Outcomes Between Eversion and Conventional Techniques in Carotid Endarterectomy
Brief Title: Comparison of Eversion and Conventional Techniques in Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, İsmail DAL, Assistant Professor Literally: Doctor Teaching Member, Kastamonu University
Other Study IDs: KastamanuU
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerosis Occlusive Disease; Stroke (CVA) or Transient Ischemic Attack; Endarterectomy, Carotid
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Endarterectomy, Carotid; Congresses as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional endarterectomy: Who were performed conventional,primarily endarterectomy patients are included this group
  Interventions: Procedure: Carotid endarterectomy, conventional
- Eversion: Who were performed eversion endarterectomy patients are included this group
  Interventions: Procedure: Carotid endarterectomy, eversion

INTERVENTIONS:
Procedure: Carotid endarterectomy, conventional — In this study, patients were divided into two groups according to whether they underwent conventional or eversion endarterectomy. Although the eversion technique is the oldest method, the conventional approach is still widely performed due to its ease of application, despite not being recommended in current guidelines. Therefore, our aim is to contribute to the literature by comparing these two methods. The conventional method is performed with a longitudinal incision extending from the common carotid artery (CCA) to the internal carotid artery (ICA) up to the end of the plaque. The arteriotomy is then closed either primarily or with the use of a patch. In our study, we performed only the primary closure method..
  Groups: Conventional endarterectomy
Procedure: Carotid endarterectomy, eversion — In this study, patients were divided into two groups according to whether they underwent conventional or eversion endarterectomy. Although the eversion technique is the oldest method, the conventional approach is still widely performed due to its ease of application, despite not being recommended in current guidelines. Therefore, our aim is to contribute to the literature by comparing these two methods.The eversion method is performed by transecting the internal carotid artery (ICA) from the common carotid artery (CCA). The arteriotomy is then closed in an end to side fashion.
  Groups: Eversion

SUMMARY:
Atherosclerotic carotid artery disease is responsible for approximately 20% of strokes worldwide, and its treatment options include medical therapy, surgery, and stenting.Surgical management is prioritized over medical and stent based approaches and can be performed using either the conventional methed closed primarily or with a patch or the eversion technique.The aim of this study was to compare the intraoperative and early postoperative outcomes of the eversion technique and the conventional method with primary closure.

ELIGIBILITY:
Inclusion Criteria:

-Patients undergoing isolated carotid endarterectomy, either emergently or electively

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients scheduled for concomitant cardiac surgery
* Reoperations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Carotid endarterectomy was performed in patients with 50-99% stenosis who had experienced stroke or transient ischemic attack (TIA) within the last six months, as well as in asymptomatic patients with 70-99% stenosis. These patients were divided into two groups according to the surgical technique applied conventional or eversion carotid endarterectomy and intraoperative and early postoperative outcomes were compared between the groups.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with stroke and death | 30 days
  All strokes and/or deaths occurring within 30 days after surgery
Number of participants with symptoms of occlusion | Postoperative 30 days
  Early carotid restenosis or occlusion within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ferguson GG, Eliasziw M, Barr HW, Clagett GP, Barnes RW, Wallace MC, Taylor DW, Haynes RB, Finan JW, Hachinski VC, Barnett HJ. The North American Symptomatic Carotid Endarterectomy Trial : surgical results in 1415 patients. Stroke. 1999 Sep;30(9):1751-8. doi: 10.1161/01.str.30.9.1751. PMID 10471419
- [Background] Wu S, Wang H, Guo J, Zhang F, Pan D, Ning Y, Gu Y, Guo L. Comparative on the effectiveness and safety of different carotid endarterectomy techniques: a single-center Retrospective Study. J Cardiothorac Surg. 2024 Jun 20;19(1):338. doi: 10.1186/s13019-024-02838-0. PMID 38902703
- [Background] Schneider JR, Helenowski IB, Jackson CR, Verta MJ, Zamor KC, Patel NH, Kim S, Hoel AW; Society for Vascular Surgery Vascular Quality Initiative and the Mid-America Vascular Study Group. A comparison of results with eversion versus conventional carotid endarterectomy from the Vascular Quality Initiative and the Mid-America Vascular Study Group. J Vasc Surg. 2015 May;61(5):1216-22. doi: 10.1016/j.jvs.2015.01.049. PMID 25925539
- [Background] Jonsson M, Lindstrom D, Wanhainen A, Djavani Gidlund K, Gillgren P. Near Infrared Spectroscopy as a Predictor for Shunt Requirement During Carotid Endarterectomy. Eur J Vasc Endovasc Surg. 2017 Jun;53(6):783-791. doi: 10.1016/j.ejvs.2017.02.033. Epub 2017 Apr 19. PMID 28431821
- [Background] Ben Ahmed S, Daniel G, Benezit M, Ribal JP, Rosset E. Eversion carotid endarterectomy without shunt: concerning 1385 consecutive cases. J Cardiovasc Surg (Torino). 2017 Aug;58(4):543-550. doi: 10.23736/S0021-9509.16.08495-0. Epub 2015 Feb 12. PMID 25673097
- [Background] Deser SB, Demirag MK, Kolbakir F. Does surgical technique influence the postoperative hemodynamic disturbances and neurological outcomes in carotid endarterectomy? Acta Chir Belg. 2019 Apr;119(2):78-82. doi: 10.1080/00015458.2018.1459364. Epub 2018 Apr 27. PMID 29701500
- [Background] Yuruk MA, Ozdemir AC. Eversion versus conventional carotid endarterectomy: A retrospective cohort study. Medicine (Baltimore). 2025 Aug 15;104(33):e43908. doi: 10.1097/MD.0000000000043908. PMID 40826780
- [Background] Yasa H, Akyuz M, Yakut N, Aslan O, Akyuz D, Ozcem B, Tulukoglu E, Gurbuz A. Comparison of two surgical techniques for carotid endarterectomy: conventional and eversion. Neurochirurgie. 2014 Feb-Apr;60(1-2):33-7. doi: 10.1016/j.neuchi.2013.12.003. Epub 2014 Mar 24. PMID 24673880
- [Background] Lee JH, Suh BY. Comparative results of conventional and eversion carotid endarterectomy. Ann Surg Treat Res. 2014 Oct;87(4):192-6. doi: 10.4174/astr.2014.87.4.192. Epub 2014 Sep 25. PMID 25317414
- [Background] Kakisis JD, Antonopoulos CN, Moulakakis KG, Schneider F, Geroulakos G, Ricco JB. Protamine Reduces Bleeding Complications without Increasing the Risk of Stroke after Carotid Endarterectomy: A Meta-analysis. Eur J Vasc Endovasc Surg. 2016 Sep;52(3):296-307. doi: 10.1016/j.ejvs.2016.05.033. Epub 2016 Jul 4. PMID 27389942
- [Background] Gahremanpour A, Perin EC, Silva G. Carotid artery stenting versus endarterectomy: a systematic review. Tex Heart Inst J. 2012;39(4):474-87. PMID 22949763